CLINICAL TRIAL: NCT06607640
Title: Study on the Association of Time Pattern of Outdoor Activity With Axial Length and Myopia of Preschool Children and Its Intervention
Brief Title: Study of the Intervention Effect of Outdoor Activity Period Patterns in Promoting Myopia Among Preschool Children
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fangbiao Tao (Other)
Responsible Party: Sponsor-Investigator, Fangbiao Tao, Professor, Anhui Medical University
Organization: Anhui Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20240666
Record Dates: First submitted 2024-09-19; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Axial Length; Myopia
MeSH Terms: conditions — Myopia | interventions — Methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: Increase outdoor activity time during specific time periods. (Experimental): The intervention group received an additional 1 hour of outdoor activity during a specific time period on each school day, with the intervention lasting for one year.
  Interventions: Behavioral: Increase outdoor activity time during specific time periods
- continued their regular indoor or outdoor routine (No Intervention): The control group continued their regular indoor or outdoor routine.

INTERVENTIONS:
Behavioral: Increase outdoor activity time during specific time periods — The specific time periods of outdoor activity found to be beneficial for myopia prevention will be used as the intervention "target," and a one-year intervention will be initiated.
  Other Names: Intervention with a specific outdoor activity model
  Arms: Intervention: Increase outdoor activity time during specific time periods.

SUMMARY:
This study is a randomized controlled trial based on outdoor activity interventions at specific time periods, involving preschool children aged 4 to 5 years. It compared the axial length and myopia incidence between the intervention group and the control group at the 6th and 12th months of the intervention to determine the effect of outdoor activities at specific time periods on the prevention of myopia in preschool children. Additionally, the study investigated the association between outdoor activities at specific time periods and axial length and myopia in preschool children.

DETAILED DESCRIPTION:
Preschool children with insufficient outdoor activity during specific time periods from one kindergarten were assigned to the intervention group, while those from another kindergarten with insufficient outdoor activity during specific time periods were assigned to the control group. The intervention group received an additional 1 hour of outdoor activity during a specific time period on each school day, while the control group did not receive any intervention and continued their regular routine. The intervention lasted for one year.

Participants underwent multiple assessments after joining the study. These assessments took place at baseline, at the 6th month of the intervention, and at the 12th month.

ELIGIBILITY:
Inclusion Criteria:

* Students and their families were informed and voluntarily participated in the study, with parents signing the informed consent form.
* Able to cooperate with eye examinations and questionnaires.

Exclusion Criteria:

* Communication barriers, unable to cooperate.
* Strabismus, amblyopia, or any other ocular or systemic diseases that may affect refractive development.
* Children currently using orthokeratology lenses or rigid contact lenses.
* Using other interventions (such as acupuncture, massage, medication, ear acupuncture, etc.) to control myopia, apart from school eye exercises.

Ages: 4 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 210 (Estimated)
Dates: Start 2024-09-21 (Estimated); Primary Completion 2025-09-21 (Estimated); Study Completion 2025-12-21 (Estimated)

PRIMARY OUTCOMES:
The changes in axial length (AL) and spherical equivalent (SE) compared to baseline after one year of intervention | at baseline, at the 6th month of the intervention, and at the 12th month.
  The ocular physiological parameters, including axial length (AL), horizontal and vertical corneal curvature (K1 and K2), were measured using an optical biometer (model IOL Master 700). Each eye was measured three times, and if the difference between any two measurements exceeded 0.05 mm, the process was repeated until the difference was less than this value.An objective examination method was used under non-cycloplegic conditions (i.e., without pupil dilation), utilizing a tabletop automatic refractometer (ISO 10342-2010 Ophthalmic Instruments - Refractometers). The spherical equivalent (SE) was calculated as follows: SE = sphere power + 1/2 cylinder power.

SECONDARY OUTCOMES:
The incidence of myopia. | at baseline, at the 6th month of the intervention, and at the 12th month.
  The incidence of myopia is defined as the occurrence of myopia in children who were not myopic at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Yang Feng, Principal Investigator — Anhui Medical University